CLINICAL TRIAL: NCT02354365
Title: Transpulmonary Pressure Monitoring as a Guide to Ventilator Management
Brief Title: Measuring Lung Pressures in Critically Ill Children Who Are on Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Christopher J. L. Newth, MD, Pediatric Critical Care Medicine, Attending Physician, Children's Hospital Los Angeles
Other Study IDs: CCI-13-00370
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2023-10

CONDITIONS: Transpulmonary Pressure; Pressure.Rate Product; Guide to Mechanical Ventilator Management; Extubation Readiness
Keywords: PEEP adjustment; Tidal Volume; Driving Pressure; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal lungs: Mechanically ventilated patients without pulmonary parenchymal disease or lower airway disease as measured by flow volume loops consistent with expiratory flow obstruction (e.g. seizures, apnea, upper airway obstruction).
  Interventions: Device: Transpulmonary Pressure measurement
- Acute Hypoxic Respiratory Failure: Mechanically ventilated patients with two consecutive Saturation to FiO2 (SF) ratio < 265 or PaO2 to FiO2 (PF) ratio < 300 (e.g. pneumonia, ARDS).
  Interventions: Device: Transpulmonary Pressure measurement
- Obstructive airway disease: Mechanically ventilated patients with flow volume loops consistent with expiratory flow obstruction (e.g. asthma, bronchiolitis).
  Interventions: Device: Transpulmonary Pressure measurement

INTERVENTIONS:
Device: Transpulmonary Pressure measurement — Transpulmonary pressure measurements are done by placing a catheter (often combined with a feeding tube) into the esophagus of a patient. Intermittently, the esophageal pressure is measured by inflating a small balloon on this catheter. The resulting esophageal pressure is accepted as representing the pleural pressure. The difference between this pressure and the airway pressure is the transpulmonary pressure and PEEP is raised or lowered to make this value zero so that the forces distending the alveoli are just balanced with the natural elasticity of the lung which wants to collapse the alveoli.

SUMMARY:
Typically doctors adjust the settings on the ventilator to ensure that children receive enough help to decrease the work they perform to breathe, receive enough oxygen through the machine to pass into the blood and to the organs, and remove acid that builds up in the blood. However, sometimes the settings we choose can result in damage to the lungs. We are trying to find a better way to determine the best ventilator settings, which can minimize potential damage to the lungs, and still provide children with enough support to decrease the work they have to do to breathe. We believe we can personalize these choices for each child by looking at the pressure that is generated in the chest while children breathe with the ventilator. This is accomplished by using a small tube which goes through the nose and into the esophagus or stomach, which is hooked up to a computer or the ventilator to monitor pressure. This same tube can then also be used to monitor how much work children need to do to breathe as we are turning down the ventilator in preparation to remove the breathing tube.

DETAILED DESCRIPTION:
Any patient weighing >2 kg between the ages of > 37 weeks corrected gestational age and <18 years who is intubated and mechanically ventilated will be eligible for the study. We seek to group patients into 3 potential cohorts:

i. Normal Lungs (maximum 30 patients): Mechanically ventilated patients without pulmonary parenchymal disease or lower airway disease as measured by flow volume loops consistent with expiratory flow obstruction (e.g. seizures, apnea, upper airway obstruction). ii. AHRF (maximum 15 patients): Mechanically ventilated patients with two consecutive Saturation to FiO2 (SF) ratio < 265 or PaO2 to FiO2 (PF) ratio < 300 (e.g. pneumonia, ARDS). iii. Obstructive airway disease (15 patients): Mechanically ventilated patients with flow volume loops consistent with expiratory flow obstruction (e.g. asthma, bronchiolitis).

Patients with a corrected gestational age of < 37 weeks or above 18 years of age. Patients with esophageal pathology or inability to utilize an esophageal probe due to anatomy, those on a high frequency oscillator or jet ventilator and those with uncorrected or persistent cyanotic congenital heart diseases will be excluded. Also, patients with an endotracheal tube leak of more than 18% or inability to measure volume, pressure or flow at the endotracheal tube will be excluded from the study.

Participation of this study can last for the duration of mechanical ventilation as pulmonary measurements will be taken during the initial phase as well as during the weaning phase of mechanical ventilation. Once patients are enrolled and informed consents obtained, an esophageal catheter will be inserted and remain in place until after extubation. The available catheters (7 and 16 French) used will be similar to size of feeding tubes used for intubated patients. These catheters/feeding tubes are often used in PICU and NICUs and are FDA 510K approved. There has been published data from our PICU for the use of these catheters in the neonatal population. For neonates and younger patients 2 kg to 10 kg, we will be using the 7Fr catheters. For older patients > 10 kg, we will be using the 16 Fr catheters. Patients that are intubated and not in the study have similar sized feeding catheters (that do not have the manometer function) routinely placed by bedside nursing staff for feeding or temperature monitoring purposes. The esophageal catheters function as both a manometer as well as a feeding tube that stays in place for the duration of mechanical ventilation. The manometer part of the catheter is located at the 1/3 of the catheter while the same catheter's distal port that serves as a feeding tube projects into the stomach. We will limit our placement of the esophageal catheter to three attempts per day. Once it is in optimal position, there will not be a need to re-adjust the catheter for pressure monitor or feeding purposes. The catheter will stay in place for duration of mechanical ventilation. Confirmation of the esophageal catheter placement will be made when the patient obtains a daily chest x-ray for routine clinical care. There will be no additional radiation exposure for intubated patients that are participating in this study than those that are not participating in this study . The esophageal catheter will be connected to the Avea mechanical ventilator and all parts will be check to ensure they are properly functioning. In order to facilitate TPP measurements, patients will need to be well sedated. During routine nursing care, mechanically ventilated patients either receive continuous or bolus sedation medication. We will time the TPP measurements to be done after patient has received bolus sedation medication.

Baseline ventilator settings will be collected. At patients' baseline ventilator settings, cardiac output (CO) will be measured using an ultrasound cardiac output monitor (USCOM). TPP measurements will be obtained at PEEP while performing an expiratory hold on the ventilator. TPP will then be obtained at PIP while performing and inspiratory hold on the ventilator. Once TPP measurements completed, PEEP will be adjusted by 2cm H2O increments to TPP. For every 2cm H2O adjustment on the ventilator, we will observe for patient tolerance of ventilator change for 2 minutes. If patients show any signs of intolerance (decrease SpO2 > 5%, increase in end tidal CO2 by more than 10 torr, heart rate >40 bpm from baseline, clinical respiratory distress), ventilator settings will be returned to baseline. Once PEEP has been adjusted to TPP, CO will be measured again using the USCOM. Measurements (CO, TPP at PEEP, TPP at PIP) will be done three times to ensure reproducibility and an average measurement of the three will be used for data description. TPP measurements will be done daily for up to 7 days. We will discontinue TPP measurements once patients are recovering and entering the weaning phase of mechanical ventilation (this is clinically determined by the primary care team in the PICU). The average length of mechanical ventilation for children in the PICU is 5-6 days, therefore an estimate of the number of TPP measurements will be 5-6 measurements.

For the later part of the study, when patients are consistently breathing spontaneously and have entered the weaning phase of ventilation, the same esophageal catheter used in the first part of the study will be used to measure pressure rate product as a surrogate for work of breathing while patients are trialed on minimal ventilator support. The esophageal catheter will be connected to the Bicore, a device that will monitor pulmonary measurements using the esophageal catheter to obtain pressure rate product measurements. The PRP will be measured with each decrease in setting of minimal ventilator support (starting from pressure support/PEEP of 10/5 cm H20 to 5/5 cm H20 to CPAP of 5cm H20). Patients will be placed on each setting for a 5 minute period and monitored for any signs of intolerance (decrease SpO2 > 5%, increase in end tidal CO2 by more than 10 torr, heart rate >40 bpm from baseline, clinical respiratory distress). Should patients not tolerate the decrease in settings of support, ventilator settings will be returned to baseline prior to changes made.

Analysis will be largely descriptive and provide information for the development of a transpulmonary pressure based protocol for ventilator management. Specifically, we will examine typical differences between PEEP set by clinicians, those recommended by available PEEP/FiO2 titration tables (ARDSNET 2000) and those recommended based on transpulmonary pressure, to determine whether there would be potential differences in choice of PEEP based on the method chosen. We will use the data to explore decision points for peak inspiratory pressure, again comparing differences between airway pressure and alveolar pressure, particularly as PEEP is changed. Finally, for aim 2, we seek to determine the potential decrease in number of days of mechanical ventilation if a minimum effort of breathing was used for the determination of extubation readiness. This will inform power calculations for future studies in which we may consider this endpoint, rather than actual extubation.

ELIGIBILITY:
Inclusion Criteria:

We seek to group patients into 3 potential cohorts:

* Normal Lungs (maximum 30 patients): Mechanically ventilated patients without pulmonary parenchymal disease or lower airway disease as measured by flow volume loops consistent with expiratory flow obstruction (e.g. seizures, apnea, upper airway obstruction).
* AHRF (maximum 15 patients): Mechanically ventilated patients with two consecutive Saturation to FiO2 (SF) ratio < 265 or PaO2 to FiO2 (PF) ratio < 300 (e.g. pneumonia, ARDS).
* Obstructive airway disease (15 patients): Mechanically ventilated patients with flow volume loops consistent with expiratory flow obstruction (e.g. asthma, bronchiolitis)

Exclusion Criteria:

• Patients with a corrected gestational age of < 37 weeks or above 18 years of age. Patients with esophageal pathology or inability to utilize an esophageal probe due to anatomy, those on a high frequency oscillator or jet ventilator and those with uncorrected or persistent cyanotic congenital heart diseases will be excluded. Also, patients with an endotracheal tube leak of more than 18% or inability to measure volume, pressure or flow at the endotracheal tube will be excluded from the study

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any patient weighing >2 kg between the ages of > 37 weeks corrected gestational age and <18 years who is intubated and mechanically ventilated in the pediatric intensive care unit at Children's Hospital Los Angeles will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary pressure | Two years
  Effect of cardiac index of increasing PEEP guided by transpulmonary pressure at PEEP.

SECONDARY OUTCOMES:
Pressure rate product (PRP) | Two years
  Effect on PRP as measure of effort of breathing while weaning on PEEP guided by transpulmonary pressure at PEEP

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Newth, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ingaramo OA, Ngo T, Khemani RG, Newth CJ. Impact of positive end-expiratory pressure on cardiac index measured by ultrasound cardiac output monitor*. Pediatr Crit Care Med. 2014 Jan;15(1):15-20. doi: 10.1097/PCC.0b013e3182976251. PMID 24389709
- [Background] Ross PA, Khemani RG, Rubin SS, Bhalla AK, Newth CJ. Elevated positive end-expiratory pressure decreases cardiac index in a rhesus monkey model. Front Pediatr. 2014 Dec 3;2:134. doi: 10.3389/fped.2014.00134. eCollection 2014. PMID 25520944
- [Background] Hotz JC, Sodetani CT, Van Steenbergen J, Khemani RG, Deakers TW, Newth CJ. Measurements Obtained From Esophageal Balloon Catheters Are Affected by the Esophageal Balloon Filling Volume in Children With ARDS. Respir Care. 2018 Feb;63(2):177-186. doi: 10.4187/respcare.05685. Epub 2017 Oct 31. PMID 29089460
- [Result] Virk MK, Hotz JC, Wong W, Khemani RG, Newth CJL, Ross PA. Minimal Change in Cardiac Index With Increasing PEEP in Pediatric Acute Respiratory Distress Syndrome. Front Pediatr. 2019 Jan 29;7:9. doi: 10.3389/fped.2019.00009. eCollection 2019. PMID 30761278